CLINICAL TRIAL: NCT05684588
Title: Post-COVID-19 Sequelae: Osteonecrosis of Femoral Head
Acronym: Covid-ON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FROM- O- Covid-ON - 2021
Record Dates: First submitted 2021-11-11; First posted 2023-01-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Osteonecrosis
Keywords: Femoral osteonecrosis; Corticosteroids; COVID-19
MeSH Terms: conditions — Osteonecrosis; COVID-19 | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: This is an experimental (non-pharmacological) diagnostic, pilot and monocentric study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Instrumental diagnostic evaluation (Other): After enrollment all patients will undergo an instrumental evaluation including a radiography (according to clinical practice) and a magnetic resonance (experimental procedure outside clinical practice), at 1 year from previous hospitalization
  Interventions: Diagnostic Test: Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance — After enrollment a Magnetic Resonance without medium contrast, at 1 year from previous hospitalization

SUMMARY:
During the most recent pandemy COVID-19, various advises concerning complications following high corticosteroid doses administration were pubblished in 2020.

However, evidence is lacking about the incidence of Non-traumatic osteonecrosis of the femoral head (ONFH) in patients experiencing COVID-19. The aim of the present proposal is to obtain a quantitative estimation of ONFH cases among patients previoulsy hospitalized and treated for COVID-19 at ASST-Papa Giovanni XXIII.

DETAILED DESCRIPTION:
Non-traumatic osteonecrosis of the femoral head (ONFH) is usually asimptomatic, but in advanced stages involves disabilities, leading to the lost of the joint functions.

The classification of the osteonecrosis type is based on clinical and radiographical criteria. Among these, the magnetic resonance (RM) plays a crucial role for detecting lesions in the early asymptomatic phase.

An high incidence of ONFH has been described during the SARS-1 pandemy: it was observed that 40% of males younger than 60, under treatment with corticosteroids, experienced it.

Based on these evidences and avises concerning complications caused by intensive corticosteroid therapy during 2020, the investigators have hypothesized that the ONFH could be underestimated in patients affected by COVID-19 and that it would be diagnosed only in its advanced disabling phase. Therefore, the main aim of this investigation is to obtain an early estimation of cases experiencing ONFH through RM as long-term sequela of COVID-19, including the assessment of articular sites involved. This will be evaluated in patients hospitalized and treated for COVID-19 at ASST-Papa Giovanni XXIII between February 23, 2020 and May 21, 2020.

After enrollment one visit and an instrumental assessment of hip status, including an RM and a radiography, will be scheduled in order to detect lesions at least at 1 year from previous hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age > 18 and < 60 years old
* Hospitalization between 23-Feb-2020 and 21-May-2020 because of COVID-19 diagnosis
* Hospitalization duration > 25 days
* Treatment with steroid drugs during hospitalization (total cumulative dose > 2 g)
* Signature of written informed consent

Exclusion Criteria:

* Presence of any implantable medical device defined as 'unsafe' for RM (eg. Cardiac pacemaker; vascular stent and gastrointestinal clips evaluated as 'unsafe')
* Previous experience with episodes and symptoms associated with claustrophobia.

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with femoral osteonecrosis | 1 year after previous hospitalization
  Number of patients showing osteonecrotic lesions

SECONDARY OUTCOMES:
Description of patients clinical features | hospitalization time 89 days
  Diseases and relevant clinical characteristic at the time of previous hospitalization for COVID-19
Description of COVID-19 | hospitalization time 89 days
  COVID-19 outcome in term of worsening (Continuous Positive Airway Pressure - CPAP use; invasive ventilation methods) and improvement status (discharge from Intensive Care Unit -ICU; discharge from hospital)
Description of therapies employed during hospitalization | hospitalization time 89 days
  Description of therapies including oxygen based therapy, oral anticoagulants (TAO), steroid drugs and other
Definition of the stage of ONFH cases | 1 year after previous hospitalization
  Stage of ONFH is defined according to ARCO classification criteria
Number of all ON types that will be detected | 1 year after previous hospitalization
  ON detected in other anatomical sites will be described including proximal humerus and knee
To describe and define the stage of all ON cases | 1 year after previous hospitalization
  Stage of other ON types as assessed by ARCO classification criteria

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ca Castelli, Prof, Study Chair — FROM-Fondazione per la Ricerca Ospedale di Bergamo
Locations (1):
- ASST-Papa Giovanni XXIII, Bergamo, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No